CLINICAL TRIAL: NCT01363492
Title: An Open-Label Clinical Trial of Replagal® Enzyme Replacement Therapy in Children With Fabry Disease Who Are Naive to Enzyme Replacement Therapy
Brief Title: Safety Study of Replagal® Therapy in Children With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-REP-084
Record Dates: First submitted 2011-03-31; First posted 2011-06-01 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
Keywords: agalsidase alfa; Replagal; Enzyme Replacement Therapy
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Replagal 0.2 mg/kg every other week (EOW) (Experimental)
  Interventions: Biological: Replagal (agalsidase alfa)

INTERVENTIONS:
Biological: Replagal (agalsidase alfa) — 0.2 mg/kg administered over 40 minutes every other week (EOW)
  Other Names: agalsidase alfa

SUMMARY:
The purpose of this study is to assess the safety of Replagal in children with Fabry disease who who have not previously been treated with enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
In 2008, a change in the agalsidase alfa drug substance manufacturing process was made. There are no changes to the drug product formulation, manufacturing site, manufacturing process, or container closure.

An agalsidase alfa bioreactor manufacturing process (agalAF1) utilizing animal component-free media replaced the previous roller bottle (RB) process.

This study will evaluate the safety of Replagal AF, manufactured using the new bioreactor process at a dose of 0.2 mg/kg infused IV over 40 minutes, every other week (EOW) in children with Fabry disease who are 7 years to less than 18 years of age and who are naive to ERT.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled in this study.

1. All patients must be diagnosed with Fabry disease by the following criteria:

   * Male Patients: The patient is a hemizygous male with Fabry disease as confirmed by a deficiency of alfa-galactosidase A activity measured in serum, leukocytes, or fibroblasts or has a confirmed mutation of the alfa-galactosidase-A gene.
   * Female Patients: The patient is a heterozygous female with Fabry disease as confirmed by a mutation of the alfa-galactosidase A gene.

   Note: If the diagnosis of Fabry disease is previously documented in the patient's medical record, screening tests do not need to be repeated.
2. The patient is 7 to <18 years of age
3. The patient is ERT-naïve
4. Adequate general health (as determined by the Investigators) to undergo the specified phlebotomy regimen and protocol-related procedures and no safety or medical contraindications for participation
5. The minor child must assent to participate in the protocol and the parent(s) or legally authorized representative(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed with the child and the child's parent(s) or legally authorized representative(s)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Patient and/or the patient's parent(s) or legally authorized representative(s) are unable to understand the nature, scope, and possible consequences of the study
2. Patient is unable to comply with the protocol, eg, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for evaluations, or is otherwise unlikely to complete the study, as determined by the Investigator or the medical monitor.
3. Otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-05-12 (Actual); Primary Completion 2013-04-17 (Actual); Study Completion 2013-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Emory Division of Medical Genetics, Decatur, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - O & O Alpan LLC, Fairfax, Virginia

REFERENCES:
- [Derived] Goker-Alpan O, Longo N, McDonald M, Shankar SP, Schiffmann R, Chang P, Shen Y, Pano A. An open-label clinical trial of agalsidase alfa enzyme replacement therapy in children with Fabry disease who are naive to enzyme replacement therapy. Drug Des Devel Ther. 2016 May 25;10:1771-81. doi: 10.2147/DDDT.S102761. eCollection 2016. PMID 27307708

RESULTS

PARTICIPANT FLOW:
Groups:
- Replagal® (0.2 mg/kg): 0.2 mg/kg Replagal (agalsidase alfa) administered over 40 minutes every other week (EOW)
Period: Overall Study
Arm/Group | Replagal® (0.2 mg/kg)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Replagal (0.2 mg/kg): 0.2 mg/kg Replagal (agalsidase alfa) administered over 40 minutes EOW
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.16 (2.992)
Age, Customized [Count of Participants; unit: Participants] — Age at informed consent
  Participants
    <=18 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 14
Heart rate variability parameter SDNN [Mean (Standard Deviation); unit: msec] | 103.46 (32.928)
Heart rate variability parameter rMSSD [Mean (Standard Deviation); unit: msec] | 75.92 (45.747)
Heart rate variability parameter pNN50 [Mean (Standard Deviation); unit: msec] | 32.79 (19.997)
Left Ventricular Mass Index (LVMI) [Mean (Standard Deviation); unit: (g/m^2.7)] | 35.37 (10.129)
Midwall Fractional Shortening (MFS) [Mean (Standard Deviation); unit: (%)] | 18.63 (2.891)
Plasma Gb3 [Mean (Standard Deviation); unit: (nmol/mL)] | 14.79 (12.228)
Urine Gb3 [Mean (Standard Deviation); unit: (nmol/g creatinine)] | 1775.08 (3691.087)

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Event (SAE)
Time Frame: Baseline to week 55
Measure: Number; unit: events
Groups:
- Replagal (0.2 mg/kg): 0.2 mg/kg Replagal (agalsidase alfa) administered over 40 minutes every other week (EOW)
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
events | 0

2. Primary Outcome: Number of Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline to week 55
Measure: Number; unit: events
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
events | 166

3. Primary Outcome: Development of IgG Anti-Agalsidase Alfa Antibody
Description: Reflects development of Anti-Agalsidase antibodies post baseline
Time Frame: Baseline to Week 55
Measure: Number; unit: participants
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
participants | 1

4. Secondary Outcome: Change From Baseline in LVMI
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: (g/m^2.7)
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
(g/m^2.7) | 0.16 (6.059)

5. Secondary Outcome: Change From Baseline in MFS
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
(%) | -0.62 (3.596)

6. Secondary Outcome: Change From Baseline in Plasma Gb3
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: (nmol/mL)
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 14
(nmol/mL) | -5.71 (8.799)

7. Secondary Outcome: Change From Baseline in Urine Gb3
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: (nmol/g creatinine)
Arm/Group | Replagal (0.2 mg/kg)
Number analyzed (Participants) | 12
(nmol/g creatinine) | -1403.25 (3636.711)

8. Primary Outcome: Change From Baseline in Heart Rate Variability Parameter SDNN
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Replagal 0.2 mg/kg: 0.2 mg/kg Replagal (agalsidase alfa) administered over 40 minutes EOW
Arm/Group | Replagal 0.2 mg/kg
Number analyzed (Participants) | 13
msec | 10.46 (24.223)

9. Primary Outcome: Change From Baseline in Heart Rate Variability Parameter rMSSD
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Replagal 0.2 mg/kg
Number analyzed (Participants) | 13
msec | 1.46 (53.502)

10. Primary Outcome: Change From Baseline in Heart Rate Variability Parameter pNN50
Time Frame: Baseline to week 55
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Replagal 0.2 mg/kg
Number analyzed (Participants) | 13
msec | -4.13 (20.166)

ADVERSE EVENTS:
Time Frame: Baseline to week 55
Groups:
- Replagal® (0.2 mg/kg): 0.2 mg/kg Replagal (agalsidase alfa) administered over 40 minutes EOW
Arm/Group | Replagal® (0.2 mg/kg)
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal® (0.2 mg/kg) (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hordeolum (Eye disorders) | 1 (1)
Retinal vascular disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (12)
Tooth malformation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (12)
Chest discomfort (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 6 (8)
Seasonal allergy (Immune system disorders) | 1 (1)
Alveolar osteitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (4)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Liver palpable subcostal (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (7)
Paraesthesia (Nervous system disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication